CLINICAL TRIAL: NCT06063460
Title: Investigation of Halitosis, Taste and Smell in Terms of Periodontal Condition Stated by Patients and Periodontal Diagnosis by Dentists, and Then Evaluation of Change Before and After Treatment
Brief Title: The Impact of Non-surgical Periodontal Therapy on Patients' Halitosis, Taste Perception, and Smell Sensation
Status: Enrolling by invitation | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, Assistant professor, Necmettin Erbakan University
Other Study IDs: PerioSmellTaste
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis | interventions — Smell; Taste

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ginigival health: The VAS scale will be filled about halitosis, smell and taste perception by patients diagnosed with gingival health during the exam.Patients will be called for a follow-up check in the 1st and 3rd months. Periodontal examinations will be repeated. The VAS scale will be filled in again with halitosis, smell and taste perception.
  Interventions: Diagnostic Test: Periodontal examination; Other: baseline questionnaire about sociodemographic characteristics, smoking habits, oral hygiene habits, halitosis, smell and taste perception; Other: 1. month periodontal evaluation and repeat questionnaire; Other: 3. month periodontal evaluation and repeat questionnaire
- Gingivitis: Patients diagnosed with gingivitis during will have the VAS scale filled in with halitosis, smell and taste perception. Phase 1 treatment will be applied. Patients will be called for a follow-up check in the 1st and 3rd months. Periodontal examinations will be repeated. The VAS scale will be filled in again with halitosis, smell and taste perception.
  Interventions: Diagnostic Test: Periodontal examination; Other: baseline questionnaire about sociodemographic characteristics, smoking habits, oral hygiene habits, halitosis, smell and taste perception; Other: phase I periodontal treatment; Other: 1. month periodontal evaluation and repeat questionnaire; Other: 3. month periodontal evaluation and repeat questionnaire
- Periodontitis: Patients diagnosed with periodontitis d will have the VAS scale filled in with halitosis, smell and taste perception. Phase 1 treatment will be applied. Patients will be called for a follow-up check in the 1st and 3rd months. Periodontal examinations will be repeated. The VAS scale will be filled in again with halitosis, smell and taste perception.
  Interventions: Diagnostic Test: Periodontal examination; Other: baseline questionnaire about sociodemographic characteristics, smoking habits, oral hygiene habits, halitosis, smell and taste perception; Other: phase I periodontal treatment; Other: 1. month periodontal evaluation and repeat questionnaire; Other: 3. month periodontal evaluation and repeat questionnaire

INTERVENTIONS:
Diagnostic Test: Periodontal examination — Periodontal Examination Routine In routine periodontal examination, measurements of plaque score, gingival score, pocket depths, and attachment loss will be utilized.
Other: baseline questionnaire about sociodemographic characteristics, smoking habits, oral hygiene habits, halitosis, smell and taste perception — Each patient participating in the study will complete a questionnaire detailing their age, gender, height, weight, smoking status, frequency of dental brushing, diabetes status, total annual household income, and Covid-19 history. In addition, a visual analogue scale and self-reported periodontal status questionnaire will be completed.
  Personal Periodontal Condition Questionnaire This questionnaire comprises of eight questions regarding the participants' periodontal condition.
  Graphical Analog Scale Patients were asked to rate their perception of taste, smell, and bad breath between 0 and 100 on this scale. Sense of smell (0-I cannot smell at all, 100-I can smell perfectly), sense of taste (0-I cannot taste at all, 100-I can smell perfectly), mouth. The odor will be graded from 0 (no bad breath) to 100 (extremely awful breath).
Other: phase I periodontal treatment — Phase I periodontal treatment will be applied by same expert.
  Groups: Gingivitis; Periodontitis
Other: 1. month periodontal evaluation and repeat questionnaire — Periodontal examination will be performed in the 1st month, filling the questionnaire about halitosis, smell and taste perception.
Other: 3. month periodontal evaluation and repeat questionnaire — Periodontal examination will be performed in the 3rd month, filling the questionnaire about halitosis, smell and taste perception.

SUMMARY:
The goal of this observational study is to evaluate the effect of non-surgical periodontal treatment on patient halitosis, smell, and taste perception in gingivitis and periodontitis patients. The main questions it aims to answer are:

* Do gingivitis, periodontitis, and gingival health affect the patient's halitosis, taste, and smell perception?
* Does non-surgical treatment affect the patient's bad breath, perception of taste and smell? Participants will be informed about the study. No additional intervention will be performed for the study, and patients will continue their routine periodontal treatments.

DETAILED DESCRIPTION:
This research will involve 180 individuals aged 18 to 65 who applied to the Department of Periodontology at the Faculty of Dentistry at Necmettin Erbakan University for various reasons. The investigation is scheduled for September to December of 2023. After clinical and radiological evaluation, each patient diagnosed with periodontal disease in the Department of Periodontics receives initial phase-1 treatment.

Individual preference If patients who seek periodontal treatment at the Periodontology Clinic Secretariat meet the study's inclusion criteria, they will be included in the study if they agree to fill out sociodemographic information such as age, gender, education level, a visual analog scale, and a self-reported periodontal status survey prior to treatment and sign the consent form. In the investigation, participants will be diagnosed with periodontium that is clinically healthy, gingivitis, and periodontitis.

Our research is a prospective survey investigation. In the study, researchers will ask patients undergoing routine periodontal examinations in the clinic and for whom treatment is planned to complete questionnaires beforehand. Tracking of survey responses will continue until the total number of respondents has been reached. Patients will resume their routine phase 1 treatment after completing the questionnaires.

Periodontal Examination Routine In routine periodontal examination, measurements of plaque score, gingival score, pocket depths, and attachment loss will be utilized. Plaque accumulation; According to the PI defined by Silness and Löe, 0: no plaque; 1: plaque at the end of the probe; 2: plaque visible to the naked eye; 3: will be evaluated as excessive plaque accumulation. Gingival index: According to Loe and Silness, 0 indicates healthy gingiva; 1 indicates mild inflammation and discoloration, with no bleeding on probing; 2 indicates moderate inflammation, hyperemia, and bleeding on probing; and 3 indicates severe inflammation, hyperemia, ulceration, edema, and spontaneous bleeding.

Patients will be treated in accordance with the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Clinical gingival health will be defined as a probing depth of less than 3 mm and a bleeding area of less than 10%. Periodontitis will be diagnosed if interdental clinical attachment loss (CAL) is detected in 2 nonadjacent teeth or if more than 3 mm of buccal or oral CAL is detected in 2 teeth with a probing depth of 3 mm. The severity of periodontitis will be determined using a system of stages and grades. The interdental CAL at the site of the greatest loss will be used to define the four stages. Stage is used to categorize the severity and complexity of periodontitis (Stage I-II-III-IV), while grade is used to estimate the likelihood of case progression (Grades A and B).

At six sites per tooth, the probing profundity and CAL will be evaluated. For PD measurement with a periodontal probe, the probe is positioned parallel to the vertical axis of the tooth to reach the deepest point of the pocket, and the distance between the base of the pocket and the gingival margin is manually measured to the nearest millimeter mark. Similarly, CAL will be measured and manually recorded as the distance between the cementoenamel border and the bottom of the compartment. When measuring CAL, areas where the enamel-cement border is not visible will be identified through tactile sense.

Each patient participating in the study will complete a questionnaire detailing their age, gender, height, weight, smoking status, frequency of dental brushing, diabetes status, total annual household income, and COVID-19 history. In addition, a visual analog scale and self-reported periodontal status questionnaire will be completed.

Personal Periodontal Condition Questionnaire This questionnaire comprises eight questions regarding the participants' periodontal condition.

Graphical Analog Scale Patients were asked to rate their perception of taste, smell, and bad breath between 0 and 100 on this scale. Sense of smell (0-I cannot smell at all, 100-I can smell perfectly), sense of taste (0-I cannot taste at all, 100-I can smell perfectly), mouth. The odor will be graded from 0 (no bad breath) to 100 (extremely awful breath).

Statistical examination According to the results of the power analysis for the Correlation: Bivariate Normal Model performed with the G Power program (G * Power 3.1 software; Heinrich Heine University, Düsseldorf, Germany), with (margin of error) = 0.05, at a power of 0.90 (1- It was determined that 180 samples were sufficient if the ) critical correlation value was 0.3. Nonetheless, presuming 20% of patients quit, the study is expected to include a total of 216 participants.

Using the SPSS 11.0 statistical software (SPSS Inc., Chicago, IL, USA), data will be analyzed. The chi-square test will be used to investigate the relationships between qualitative variables, the t-test will be used to compare two groups in terms of quantitative variables, and one-way ANOVA will be used to determine the significance of the relationships. ANOVA will be used to compare quantitative variables between more than two groups. The relationship between qualitative variables will be analyzed using Pearson correlation. A P value of 0.05 will indicate statistical significance. The effects of sibling size, birth order, and socioeconomic status on the risk of tooth loss and periodontal disease will be evaluated and potential confounders will be controlled for using logistic regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 18-65
* Healthy periodontium, getting diagnosed with gingivitis or periodontitis

Exclusion Criteria:

* Not agreeing to participate in the study
* Having a psychiatric, mental or physical disability
* Having received periodontal treatment in the last 6 months
* Being pregnant and lactating
* Any antibiotics that may affect periodontal tissues for any reason in the last 6 months
* Having used an anti-inflammatory or other medication

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study will include 216 people aged 18-65 who applied to Necmettin Erbakan University Faculty of Dentistry Department of Periodontology for various reasons. The investigation is scheduled for July-September 2023. After clinical and radiographic evaluation, all periodontal disease patients get phase-1 treatment in the Department of Periodontics. Patients who meet the inclusion criteria and sign the consent form will be included in the study if they fill out sociodemographic information like age, gender, education level, visual analogue scale, and self-reported periodontal status survey before treatment at the Periodontology Clinic Secretariat. The study will diagnose clinically healthy periodontium, gingivitis, and periodontitis.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference between halitosis, smell and taste perception measured by VAS scale in gingival health, gingivitis and periodontitis groups at baseline | Baseline
  The senses of taste and smell were collected using a visual analogue scale (VAS), where the participants were asked to rate their ability to taste or smell. The value zero represented "no taste" or "no smell," and 100 described "excellent taste" or "excellent smell" .
  Halitosis was considered the mediator and was measured using a VAS, where the participants were asked to rate their breath odor. The scale went from a value of zero, corresponding to "no bad breath," to 100, corresponding to "extremely bad breath". 3 groups will be compared to each other.
Comparison of halitosis taste and smell perception measured by VAS scale in gingivitis and periodontitis groups, at baseline and 1 month after initial treatment | 1st month
  At the 1st month after the initial treatment, the halitosis, taste and smell perceptions of the participants in all groups will be measured with the VAS scale. The initial and 1st month results of the groups will be compared with each other. The senses of taste and smell were collected using a visual analogue scale (VAS), where the participants were asked to rate their ability to taste or smell. The value zero represented "no taste" or "no smell," and 100 described "excellent taste" or "excellent smell" .
  Halitosis was considered the mediator and was measured using a VAS, where the participants were asked to rate their breath odor. The scale went from a value of zero, corresponding to "no bad breath," to 100, corresponding to "extremely bad breath".
Comparison of halitosis taste and smell perception measured by VAS scale in gingivitis and periodontitis groups, at baseline and 3 month after initial treatment | 3rd month
  At the 3rd month after the initial treatment, the halitosis, taste and smell perceptions of the participants in all groups will be measured with the VAS scale. The initial and 1st month results of the groups will be compared with each other. The senses of taste and smell were collected using a visual analogue scale (VAS), where the participants were asked to rate their ability to taste or smell. The value zero represented "no taste" or "no smell," and 100 described "excellent taste" or "excellent smell" .
  Halitosis was considered the mediator and was measured using a VAS, where the participants were asked to rate their breath odor. The scale went from a value of zero, corresponding to "no bad breath," to 100, corresponding to "extremely bad breath".

CONTACTS AND LOCATIONS:
Overall Officials: zeynep taştan eroğlu, Study Director — Necmettin Erbakan University
Locations (1):
- Zeynep Taştan Eroğlu, Konya, Meram, Turkey (Türkiye)

REFERENCES:
- [Derived] Tastan Eroglu Z, Kalender ME, Ucan Yarkac F, Babayigit O, Ozkan Sen D. Impact of non-surgical periodontal therapy on self-perceived halitosis, and the senses of smell and taste: a prospective clinical study. BMC Oral Health. 2025 Feb 28;25(1):321. doi: 10.1186/s12903-025-05702-2. PMID 40022178